CLINICAL TRIAL: NCT01350947
Title: A Phase II Study of the Efficacy, Safety and Determinants of Response to 5-Azacitidine (Vidaza®) in Patients With Chronic Myelomonocytic Leukemia (CMML)
Brief Title: A Study of 5-Azacitidine (Vidaza®) in Patients With Chronic Myelomonocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI47081
Record Dates: First submitted 2011-04-29; First posted 2011-05-10 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Myelomonocytic Leukemia
Keywords: Chronic Myelomonocytic Leukemia; CMML
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Drug: 5-Azacitidine

INTERVENTIONS:
Drug: 5-Azacitidine — Administered on Days 1-7 of each Cycle.
  Subcutaneous administration:
  To provide a homogeneous suspension, the contents of the syringe must be re-suspended by inverting the syringe 2-3 times and vigorously rolling the syringe between the palms for 30 seconds immediately prior to administration.
  The 5-azacitidine suspension is administered subcutaneously.
  Intravenous Administration:
  5-Azacitidine solution is administered intravenously. Administer the total dose over a period of 10-40 minutes.
  Other Names: Vidaza®

SUMMARY:
The primary objective of this study is:

Response to treatment will be evaluated according to the revised International Working Group (IWG) categories natural history, hematologic improvement and cytogenetic response1;2. The primary objective is:

To determine the rate of complete hematologic response and hematologic improvement (according to IWG 2006 criteria) in CMML patients treated with 5-azacitidine.

DETAILED DESCRIPTION:
In this study, eligible patients with a confirmed diagnosis of CMML will be treated with 5-azacitidine to determine the rates of complete hematologic response, hematologic improvement, complete and partial cytogenetic response, and overall and progression free survival.

To develop biomarkers associated with response and gain insights into the mechanisms that determine response, gene expression profiling, genome-wide SNP array analysis, microRNA analysis, and DNA methylation analysis will be performed prior to therapy and at defined time points during the study. Phosphoproteomics profiling may be included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CMML as defined by the WHO criteria

   1. Persistent peripheral blood monocytosis of more than 1 x 109/L for at least 3 months and
   2. No Philadelphia chromosome or BCR-ABL fusion gene and
   3. Less than 20% blasts in the blood or bone marrow and
   4. Dysplasia in one or more of the myeloid lineages* * In the absence of dysplasia in one or more of the myeloid lineages, the diagnosis of CMML can still be made if a) - c) are met AND an acquired clonal chromosomal abnormality is present in the bone marrow cells, the monocytosis has been present for more than 3months AND all other causes of monocytosis have been ruled out.
2. Age of 18 years or older. Both men and women and members of all races and ethnic groups will be included.
3. ECOG performance status <3
4. Adequate organ function defined as:

   1. Total bilirubin <2.5 x upper limit of normal (ULN)
   2. Direct bilirubin <2 x ULN
   3. Creatinine <2 mg/dL
   4. ALT and AST <2.5 x ULN
5. Ability to understand and the willingness to sign a written informed consent document
6. Willingness to use adequate contraception for the duration of the study

Exclusion Criteria:

1. Progression to acute myeloid leukemia (defined by at least 20% blasts in the blood or bone marrow). In the unlikely event that progression to acute leukemia is demonstrated in the "screening" bone marrow biopsy, it is at the discretion of the investigator to enroll the patient after adequate discussion of the findings and alternative therapies. Enrollment of such a patient must be reported to the HCI PI.
2. Presence of activating mutations of the platelet derived growth factor receptors alpha or beta, which would suggest likely benefit from imatinib treatment (these mutations will usually be obvious from karyotyping and fluorescence in situ hybridization studies)
3. Known or suspected hypersensitivity to 5-azacitidine or mannitol
4. Clinically significant heart disease (New York Heart Association Class III or IV) or other serious intercurrent illnesses or psychiatric illness/social situations that would limit compliance with study requirements
5. Major surgery within 28 days before registration (exception: central venous line placement), or lack of full recovery from prior major surgery
6. Prior therapy with a hypomethylating agent
7. Cytotoxic chemotherapy less than 2 weeks prior to starting study medication (exception: hydroxyurea and/or anagrelide)
8. Erythropoietin or darbepoietin, G-CSF, GM-CSF, thalidomide or lenalidomide less than 2 weeks from day 1 of cycle 1
9. Concomitant cytotoxic chemotherapy (exception: hydroxyurea for up to 1 week per cycle)
10. Concomitant therapy with other investigational agents
11. Other active malignancies except basal cell carcinoma of the skin and carcinoma in situ of the cervix.
12. Pregnancy or breastfeeding (possible risk to the fetus or infant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Deininger, MD, Principal Investigator — University of Utah
Locations (3):
- United States (3):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - 5-Azacitidine: All participants enrolled.
  5-Azacitidine: Administered on Days 1-7 of each Cycle.
  Subcutaneous administration:
  To provide a homogeneous suspension, the contents of the syringe must be re-suspended by inverting the syringe 2-3 times and vigorously rolling the syringe between the palms for 30 seconds immediately prior to administration.
  The 5-azacitidine suspension is administered subcutaneously.
  Intravenous Administration:
  5-Azacitidine solution is administered intravenously. Administer the total dose over a period of 10-40 minutes.
Period: Overall Study
Arm/Group | Arm 1 - 5-Azacitidine
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All participants enrolled.
  5-Azacitidine: Administered on Days 1-7 of each Cycle.
  Subcutaneous administration:
  To provide a homogeneous suspension, the contents of the syringe must be re-suspended by inverting the syringe 2-3 times and vigorously rolling the syringe between the palms for 30 seconds immediately prior to administration.
  The 5-azacitidine suspension is administered subcutaneously.
  Intravenous Administration:
  5-Azacitidine solution is administered intravenously. Administer the total dose over a period of 10-40 minutes.
Arm/Group | All Patients
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 69 [56 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete Hematologic Response (According to IWG 2006 Criteria) in CMML Patients Treated With 5-azacitidine.
Description: Complete Hematologic Response is defined as: bone marrow evaluation shows <= 5% myeloblasts with normal maturation of all cells lines; peripheral blood evaluation shows hemoglobin >= 11 g/dL, neutrophils >= 1000/mL, platelets >= 100,000/mL, 0% blasts
Time Frame: 24 months
Measure: Number; unit: percentage of patients
Arm/Group | Arm 1 - 5-Azacitidine
Number analyzed (Participants) | 11
percentage of patients | 27

ADVERSE EVENTS:
Arm/Group | Arm 1 - 5-Azacitidine
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - 5-Azacitidine (N=11)
Fatigue (General disorders) | 1 (1)
leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Thrombocytopenia (Investigations) | 1 (1)
Hematochezia (Blood and lymphatic system disorders) | 1 (1)
seizure (Nervous system disorders) | 1 (1)
wound treatment (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - 5-Azacitidine (N=11)
Abdominal Cramping (Gastrointestinal disorders) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 7 (22)
ankle sprain (Injury, poisoning and procedural complications) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 2 (2)
anthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
back pain (Metabolism and nutrition disorders) | 2 (3)
Bacteremia (Infections and infestations) | 1 (1)
bloating (Gastrointestinal disorders) | 1 (1)
bloody discharge from urethra (Blood and lymphatic system disorders) | 1 (1)
bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Broken Blood Vessel of the Eye (Eye disorders) | 1 (1)
bruising (Skin and subcutaneous tissue disorders) | 4 (4)
cellulitis (Infections and infestations) | 2 (2)
chest lesion (Injury, poisoning and procedural complications) | 1 (1)
chest pain (General disorders) | 1 (1)
chills (General disorders) | 1 (1)
chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
cold sweats (General disorders) | 1 (1)
cold symptoms (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (10)
Cooler Lower Extremeties (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
decreased neutrophil (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (4)
dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
dry mouth (Gastrointestinal disorders) | 1 (1)
dry nose (General disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (4)
dyspepsia (Gastrointestinal disorders) | 1 (1)
dysphagia (Gastrointestinal disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Ecchymoses (Skin and subcutaneous tissue disorders) | 2 (3)
epigastric pain (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
erythmea (Skin and subcutaneous tissue disorders) | 1 (1)
eye irratation (Eye disorders) | 1 (1)
eye swelling (Eye disorders) | 1 (1)
face burning (Skin and subcutaneous tissue disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (4)
Fatigue (General disorders) | 5 (5)
flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
flu like symptoms (General disorders) | 2 (2)
foot edema (Musculoskeletal and connective tissue disorders) | 1 (1)
frequent urination (Renal and urinary disorders) | 1 (1)
headache (Nervous system disorders) | 2 (2)
Hematochezia (Blood and lymphatic system disorders) | 1 (1)
hematoma (Vascular disorders) | 3 (3)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hip pain (Injury, poisoning and procedural complications) | 1 (1)
Hot Flashes (Vascular disorders) | 1 (1)
hyperglycema (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
increased creatinine (Investigations) | 1 (1)
injection reaction (General disorders) | 3 (5)
insomnia (Psychiatric disorders) | 1 (1)
itching (Skin and subcutaneous tissue disorders) | 1 (1)
labyrinthitis (Ear and labyrinth disorders) | 1 (1)
laceration (Injury, poisoning and procedural complications) | 2 (3)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (2)
leucocytosis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Investigations) | 7 (26)
limited movement of limb (Musculoskeletal and connective tissue disorders) | 1 (1)
loose stool (Gastrointestinal disorders) | 1 (1)
malaise (General disorders) | 2 (2)
mouth sores (Gastrointestinal disorders) | 1 (1)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (11)
neuropathy (Nervous system disorders) | 1 (3)
neutropenia (Nervous system disorders) | 7 (59)
neutropenic fever (Blood and lymphatic system disorders) | 1 (2)
Night Sweats (General disorders) | 2 (2)
Nightmares (General disorders) | 1 (1)
Nose Sore (General disorders) | 1 (1)
Occasional palpitations (Cardiac disorders) | 1 (1)
oral herpes lesion (Gastrointestinal disorders) | 1 (1)
parovaria cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
pelvic pain (Reproductive system and breast disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
port site infection (Infections and infestations) | 1 (1)
Prostatitis (Renal and urinary disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 2 (3)
ear lesion (Ear and labyrinth disorders) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
rhinovirus (Infections and infestations) | 1 (1)
scalp lesions (Injury, poisoning and procedural complications) | 1 (1)
seizures (Nervous system disorders) | 1 (1)
shin lesion (Injury, poisoning and procedural complications) | 1 (1)
Sinus Infection (Injury, poisoning and procedural complications) | 2 (2)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
stomach pain (Gastrointestinal disorders) | 1 (1)
syncope (Nervous system disorders) | 1 (2)
tachycardia (Cardiac disorders) | 1 (1)
tendinitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Thrombocytopenia (Investigations) | 6 (40)
tooth infection (Investigations) | 1 (1)
tooth pain (Gastrointestinal disorders) | 1 (1)
torn ligament (Musculoskeletal and connective tissue disorders) | 1 (1)
tremor (Nervous system disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1)
viral conjunctivitis (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight Gain (Investigations) | 1 (1)
wound treatment (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes